CLINICAL TRIAL: NCT03050307
Title: A Randomized Double-Blind, Double-Dummy, Phase 3 Study to Evaluate the Efficacy and Safety of Oral TAK-438 20mg Compared to Lansoprazole 30mg Once- or Twice-Daily in the Treatment of Endoscopically Confirmed Gastric Ulcer Subjects With or Without Helicobacter Pylori Infection
Brief Title: Comparison of TAK-438 (Vonoprazan) to Lansoprazole in the Treatment of Gastric Ulcer Participants With or Without Helicobacter Pylori Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-438_302; U1111-1138-8706 (Other: WHO); CTR20170100 (Registry Identifier: CFDA)
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Gastric Ulcer
Keywords: Drug therapy
MeSH Terms: conditions — Stomach Ulcer | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAK-438 20 mg (Experimental): Helicobacter Pylori positive (HP+) participants: TAK-438 20 mg tablet, twice daily (BID) along with lansoprazole placebo-matching, capsule BID in addition to bismuth-containing quadruple antibiotic therapy for the first 2 weeks. Following 2 weeks of eradication therapy participants received TAK-438 20 mg QD along with lansoprazole matching placebo 30 mg, capsule QD for up to 6 weeks. HP negative (HP-) participants: TAK-438 20 mg tablet, (QD) along with lansoprazole matching placebo, 30 mg capsule QD for up to 8 weeks.
  Interventions: Drug: TAK-438; Drug: Lansoprazole Placebo; Drug: Bismuth-Containing Quadruple Therapy
- Lansoprazole 30 mg (Experimental): HP+ participants: Lansoprazole 30 mg, capsule, orally, BID and TAK-438 placebo-matching tablet, orally, BID along with bismuth-containing quadruple antibiotic therapy for first 2 weeks. Following 2 weeks participants received Lansoprazole 30 mg, capsule, orally, QD along with TAK-438 placebo-matching tablet, orally, QD for up to 6 weeks. HP- participants: Lansoprazole 30 mg, capsule, orally, QD along with TAK-438 placebo-matching tablet, orally, QD for up to 8 weeks.
  Interventions: Drug: Lansoprazole; Drug: TAK-438 Placebo; Drug: Bismuth-Containing Quadruple Therapy

INTERVENTIONS:
Drug: TAK-438 — TAK-438 tablets
  Other Names: Vonoprazan
  Arms: TAK-438 20 mg
Drug: Lansoprazole — Lansoprazole capsules
  Other Names: Prevacid
  Arms: Lansoprazole 30 mg
Drug: TAK-438 Placebo — TAK-438 placebo-matching tablets
  Arms: Lansoprazole 30 mg
Drug: Lansoprazole Placebo — Lansoprazole placebo-matching capsules
  Arms: TAK-438 20 mg
Drug: Bismuth-Containing Quadruple Therapy — 1 g Amoxicillin, 500 mg clarithromycin and 600 mg bismuth potassium citrate/bismuth tripotassium dicitrate, twice daily (BID).

SUMMARY:
The purpose of this study is to demonstrate the non-inferior efficacy of TAK-438 versus lansoprazole in the treatment of participants with gastric ulcer.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-438. TAK-438 is being tested to treat people who have stomach ulcers and also may or may not have Helicobacter pylori (HP) infection. This study will look at stomach ulcer healing and also the elimination of HP in people who take TAK-438 versus lansoprazole.

The study will enroll approximately 830 patients.

Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the participants and study doctor during the study (unless there is an urgent medical need):

* TAK-438 20 mg
* Lansoprazole 30 mg

Study treatment will depend upon the Helicobacter pylori infection status of the participant, and include bismuth-containing quadruple therapy for the first 2 weeks in H pylori infected (HP+) participants. HP+ participants will be asked to take a TAK- 438 tablet or a lansoprazole capsule twice daily in conjunction with bismuth-containing quadruple therapy for 2 weeks, followed up by a TAK-438 tablet or a lansoprazole capsule once daily for up to 6 weeks. HP- participants will be asked to take a TAK-438 tablet or a lansoprazole capsule once daily for up to 8 weeks.

This multi-center trial will be conducted in China, Korea, Taiwan, and Philippines. The overall time to participate in this study is up to 12 weeks. Participants will make multiple visits plus final visit at 2 weeks or 4 weeks after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has endoscopic evidence of active gastric ulcer(s) (i.e. mucosal defects with white coating [including cases associated with blood coagula as long as there is no active bleeding]) measuring 5 mm or larger in longest diameter within 14 days prior to randomization.

Exclusion Criteria:

1. Has received TAK-438 in a previous clinical study or as a therapeutic agent.
2. Has a history or clinical manifestations of significant central nervous system (CNS), cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urological, endocrine or hematological disease that, in the opinion of the investigator, would confound the study results or compromise participant safety.
3. Has been treated with Helicobacter pylori eradication therapy within 30 days prior to study treatment.
4. Has any gastric ulcer of >2 cm in any diameter or with >3 separate gastric ulcers in total as evident by endoscopy within 14 days prior to randomization.
5. Has a diagnosis of gastric malignancy or a gastric ulcer whose morphology suggested malignancy as evident by endoscopy within 14 days prior to randomization.
6. Is suspected of having acute gastro-duodenal mucosal lesions (AGDML) as evident by endoscopy within 14 days prior to randomization.
7. Has a linear ulcer (including a linear ulcer scar) that has been confirmed by endoscopy within 14 days prior to randomization.
8. Has active postoperative (e.g. endoscopic mucosal resection/endoscopic submucosal dissection) ulcer(s) as confirmed by endoscopy within 14 days prior to randomization.
9. Has duodenal ulcer that has been confirmed by endoscopy within 14 days prior to randomization.
10. Has ulcers for which medical therapy alone is not indicated (e.g., perforation, pyloric stenosis, duodenal stenosis, major bleeding).
11. Has undergone therapeutic upper gastrointestinal (GI) endoscopic therapy (e.g., endoscopic hemostasis or excision including biopsy) within 30 days prior to visit 1.
12. Has Zollinger-Ellison syndrome or gastric acid hypersecretion or those with a history of gastric acid hypersecretion.
13. Has undergone major surgical procedures within 30 days prior to Visit 1 or are scheduled to undergo surgical procedures that may affect gastric acid secretion (e.g., abdominal surgery, vagotomy or craniotomy).
14. Has a history of malignancy or was treated for malignancy within 5 years before the start of the visit 1 (the participant may be included in the study if he/she has cured cutaneous basal cell carcinoma or cervical carcinoma in situ).
15. Has a known acquired immunodeficiency syndrome or hepatitis infection, including hepatitis virus carriers (hepatitis B surface-antigen [HBsAg] - or hepatitis C virus (HCV)-antibody-positive) (the participant may be included in the study if he/she is HCV-viral load-RNA-negative).
16. Laboratory tests performed prior to randomization revealed any of the following abnormalities in the participant:

    1. Creatinine levels: >2 mg/dL (>177 μmol/L).
    2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST), or total bilirubin levels: > upper limit of normal (ULN).
17. Has hypersensitivity to TAK-438, proton pump inhibitors (PPIs), bismuth, clarithromycin, or amoxicillin. Skin testing may be performed according to local standard practice (for HP+ participants only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Clinical Science, Study Director — Takeda
Locations (81):
- China (53):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Yijishan hospital of Wan nan Medical college, Wuhu, Anhui
  - Beijing Chao Yang Hospital, Beijing, Beijing Municipality
  - The General Hospital of People's Armed Police Forces China, Beijing, Beijing Municipality
  - The Central Hospital of China Aerospace Corporation, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tong Ren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing,P.R., Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fuzhou General Hospital of Nanjing Military Area Command of Chinese PLA, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhangzhou Hospital, Zhangzhou, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Haikou People's Hospital, Haikou, Hainan
  - Shiyan Taihe Hospital, Shiyan, Hebei
  - The 2nd Xiangya Hospital Central South University, Changsha, Hu'nan
  - Chenzhou No.1 People's Hospital, Chenzhou, Hu'nan
  - Changsha Central Hospital, Yuhua, Hu'nan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Union Hospital of Tongji Medical College of Huazhong Science and Techology University, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Wuhan General Hospital of Guangzhou Military, Wuhan, Hubei
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Wuxi 4th People's Hospital, Wuxi, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - Jiangxi Nanchang 3rd Hospital, Nanchang, Jiangxi
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Jilin 4th People'S hospital, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Jilin central Hospital, Jilin, Jilin
  - Jilin Siping Central Hospital, Siping, Jilin
  - General Hospital of Shenyang Military Region, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia Hui
  - People's Hospital of Qinghai Province, Xining, Qinghai
  - The 2nd Hospital of Xi An Jiaotong University, Xi'an, Shan'xi
  - Ruijin Hospital, Shanghai Jiaotong Uni. School of Med., Huangpu Qu, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University Affiliated General Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Kunming Medical College, Kunming, Yun'nan
  - 1st Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
- Philippines (6):
  - Cebu Doctors University Hospital, Cebu City
  - St. Luke's Medical Center Global City, City of Taguig
  - De La Salle University Medical Center, Dasmarinas City, Cavite
  - Davao Doctors Hospital, Davao City
  - West Visayas State University Medical Center, Iloilo City
  - Philippine General Hospital, Manila
- South Korea (17):
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - The Catholic University of Korea, Bucheon St. Mary s Hospital, Bucheon-si, Gyeonggi-do
  - Hanyang Univerisy Guri Hospital, Guri-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Wonkwang University Hospital, Iksan-si, Jeollabuk-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Dong-A University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
- Taiwan (5):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: NOTE: IPD Sharing Time Frame has not been entered.
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Hou X, Wang J, Du Q, Tian D, Hu N, Liu D, Zhou F, Xie L, Gu L, Kudou K, Zhang S. Efficacy and Safety of Vonoprazan-Based Quadruple Therapy for the Eradication of Helicobacter pylori in Patients with Peptic Ulcers: A Pooled Analysis of Two Randomized, Double-Blind, Double-Dummy, Phase 3 Trials. Biol Pharm Bull. 2024;47(8):1405-1414. doi: 10.1248/bpb.b24-00011. PMID 39085080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 60 investigative sites in China, Korea, and Taiwan from 17 April 2017 to 26 May 2020.
Pre-assignment Details: Participants with a diagnosis of gastric ulcer (GU) with or without Helicobacter pylori (H. Pylori) infection were randomized in 1:1 ratio to receive TAK-438 and lansoprazole along with placebo (to keep the blind).
Period: Overall Study
Arm/Group | TAK-438 20 mg | Lansoprazole 30 mg
Started | 115 | 119
Completed | 107 | 110
Not Completed | 8 | 9
Not completed — Adverse Event | 4 | 2
Not completed — Significant Protocol Deviation | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Voluntary Withdrawal | 3 | 4
Not completed — Reason not Specified | 1 | 1

BASELINE CHARACTERISTICS:
Population: All Randomized Participants.
Groups:
- TAK-438 20 mg: Helicobacter Pylori positive (HP+) participants: TAK-438 20 mg tablet, twice daily (BID) along with lansoprazole placebo-matching, capsule BID in addition to bismuth-containing quadruple antibiotic therapy for the first 2 weeks. Following 2 weeks of eradication therapy participants received TAK-438 20 mg QD along with lansoprazole matching placebo 30 mg, capsule QD for up to 6 weeks. HP- participants: TAK-438 20 mg tablet, (QD) along with lansoprazole matching placebo, 30 mg capsule QD for up to 8 weeks.
- Total: Total of all reporting groups
Arm/Group | TAK-438 20 mg | Lansoprazole 30 mg | Total
Number analyzed (Participants) | 115 | 119 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (13.68) | 53.5 (13.37) | 53.7 (13.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 56
  Male | 86 | 92 | 178
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 114 | 119 | 233
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 65 | 71 | 136
  Korea, Republic Of | 44 | 42 | 86
  Taiwan, Province Of China | 6 | 6 | 12
Height [Mean (Standard Deviation); unit: cm] | 165.4 (7.49) | 167.1 (7.96) | 166.2 (7.76)
Weight [Mean (Standard Deviation); unit: kg] | 63.76 (10.743) | 66.83 (11.370) | 65.32 (11.149)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — BMI=weight (kg)/[height (m)^2]
  kg/m^2 | 23.25 (3.224) | 23.85 (3.255) | 23.56 (3.247)
Smoking classification [Count of Participants; unit: Participants]
  The Participant has Never Smoked | 49 | 52 | 101
  The Participant is a Current Smoker | 50 | 51 | 101
  The Participant is an Ex-smoker | 16 | 16 | 32
Consumption of Alcohol [Count of Participants; unit: Participants] — Participants were analyzed based on the number of drinks i.e., drinks every day, two days a week, two days a month and never drinks. Population: Number analyzed is the number of participants with data available for consumption of alcohol at Baseline.
  Participants
    Drinks Every Day: number analyzed (Participants) | 115 | 118 | 233
    Drinks Every Day | 9 | 6 | 15
    Drinks Two Days a Week: number analyzed (Participants) | 115 | 118 | 233
    Drinks Two Days a Week | 20 | 25 | 45
    Drinks Two Days a Month: number analyzed (Participants) | 115 | 118 | 233
    Drinks Two Days a Month | 17 | 25 | 42
    Never Drinks: number analyzed (Participants) | 115 | 118 | 233
    Never Drinks | 69 | 62 | 131
Caffeine Consumption [Count of Participants; unit: Participants]
  Yes (>5 Times per Week) | 22 | 29 | 51
  No (Never or <5 Times a Week) | 93 | 90 | 183
H pylori infection status (13C-UBT) [Count of Participants; unit: Participants] — Participants were evaluated for the H. Pylori infection by result of 13C Urea Breath Test. Participants with infection were categorized as positive. Participants without infection were categorized as negative. Population: Number analyzed is the number of participants with data available for H. pylori Infection status at Baseline.
  Participants
    Positive: number analyzed (Participants) | 114 | 119 | 233
    Positive | 85 | 89 | 174
    Negative: number analyzed (Participants) | 114 | 119 | 233
    Negative | 29 | 30 | 59
Characteristics of GUs: Location I [Count of Participants; unit: Participants] — Participants were categorized based on their location (location I) of ulcer of the stomach.
  Participants
    Cardiac Fundus | 2 | 2 | 4
    Upper Gastric Corpus | 5 | 4 | 9
    Middle Gastric Corpus | 11 | 7 | 18
    Lower Gastric Corpus | 10 | 13 | 23
    Gastric Angle | 37 | 42 | 79
    Pyloric Antral Zone | 50 | 51 | 101
Characteristics of GUs: Location II [Count of Participants; unit: Participants] — Participants were categorized based on their location (location II) of ulcer in the stomach. Population: Number analyzed is the number of participants with data available for Characteristics of GUs: Location II at Baseline.
  Participants
    Anterior Wall: number analyzed (Participants) | 108 | 113 | 221
    Anterior Wall | 26 | 20 | 46
    Lesser Curvature: number analyzed (Participants) | 108 | 113 | 221
    Lesser Curvature | 50 | 63 | 113
    Posterior Wall: number analyzed (Participants) | 108 | 113 | 221
    Posterior Wall | 19 | 15 | 34
    Greater Curvature: number analyzed (Participants) | 108 | 113 | 221
    Greater Curvature | 13 | 15 | 28
Characteristics of GUs: Number of ulcers [Mean (Standard Deviation); unit: number of ulcers] | 1.3 (0.56) | 1.2 (0.45) | 1.2 (0.51)
Characteristics of GUs: Ulcer morphology [Count of Participants; unit: Participants] — Participants were categorized based on the morphology (shape) of ulcer: circular, ellipsoidal, or other. Population: Number of participants analyzed is the number of participants with data available for ulcer morphology at Baseline.
  Participants
    Circular | 53 | 56 | 109
    Ellipsoid | 47 | 52 | 99
    Other | 15 | 11 | 26
Characteristics of GUs: Ulcer size [Count of Participants; unit: Participants] — Participants were categorized based on the size of ulcer: minuscule (<5 mm), minor (>=5 mm and <10 mm), intermediate (>=10 mm and <=20 mm), large (>20 mm and <30 mm), giant (>=30 mm). Categories with participants available for analysis are reported.
  Participants
    Miniscule (<5 mm) | 0 | 1 | 1
    Minor (≥5 mm and <10 mm) | 82 | 76 | 158
    Intermediate (≥10 mm and ≤20 mm) | 33 | 42 | 75
Time since onset of current ulcers [Median (Full Range); unit: days] — Time since onset of current ulcers is defined as time in days from enrolment up to the onset of current ulcer. Population: Number analyzed is the number of participants with data available for Time since onset of current ulcers at Baseline.
  days
    number analyzed (Participants) | 115 | 118 | 233
    (all) | 4.0 [1 to 175] | 4.0 [-14 to 366] | 4.0 [-14 to 366]
Use of NSAID or LDA (except topical use) at time of onset of ulcer [Count of Participants; unit: Participants] — Participants who used the Nonsteroidal Anti-Inflammatory Drug (NSAID) or Low-dose Aspirin (LDA) were categorized as 'YES'. Participants who did not use the NSAID were categorized as 'NO'.
  Participants
    Yes | 11 | 8 | 19
    No | 104 | 111 | 215
Type of ulcers [Count of Participants; unit: Participants] — Participants were categorized based on the type of ulcers: primary or recurrent.
  Participants
    Primary | 96 | 103 | 199
    Recurrent | 19 | 16 | 35
Time since onset of recurrent ulcers [Median (Full Range); unit: days] — Time since onset of recurrent ulcers is defined as time in days from enrolment up to the onset of previous ulcer. Population: Number analyzed is the number of participants with data available for time since onset of recurrent ulcers at Baseline.
  days
    number analyzed (Participants) | 11 | 6 | 17
    (all) | 393.0 [113 to 2409] | 408.5 [115 to 3756] | 393.0 [113 to 3756]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Endoscopically Confirmed Healing of Gastric Ulcers (GUs) at Weeks 4 or 8
Description: Endoscopic healing was defined as the disappearance of all white coats associated with GUs confirmed endoscopically.
Time Frame: Week 4 or 8
Population: Full Analysis Set (FAS) population included all randomized participants who received at least 1 dose of the study drug. Overall number of participants analyzed were participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-438 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 112 | 114
percentage of participants | 91.1 [84.193 to 95.635] | 94.7 [88.896 to 98.044]
Statistical Analysis 1: Comparison: TAK-438 20 mg vs Lansoprazole 30 mg; Test type: Non-Inferiority — If the lower bound of the 95% CI is ≥-8%, noninferiority for TAK-438 relative to lansoprazole with regard to gastric ulcer healing was declared; Exact (Clopper-Pearson) = -3.7, 95% CI 2-sided [-10.966 to 3.339]

2. Secondary Outcome: Percentage of Helicobacter Pylori Infected (HP+) Participants With Successful HP Eradication After 4 or 8 Weeks of Treatment
Description: HP infection status was determined by 13C-UBT. The urea breath test is used to detect infection with HP, a bacteria associated with stomach ulcers, by testing individual breath samples in a central laboratory. The data is provided only for HP+ participants. The participant could take 4 or 8 weeks of treatment for GU healing, then additional 4 weeks later, to have the urea breath test (UBT) test to detect HP.
Time Frame: 4 weeks post treatment (up to approximately 12 weeks)
Population: FAS population included all randomized participants who received at least 1 dose of the study drug. Overall number of participants analyzed were participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- TAK-438 20 mg: Helicobacter Pylori positive (HP+) participants: TAK-438 20 mg tablet, twice daily (BID) along with lansoprazole placebo-matching, capsule BID in addition to bismuth-containing quadruple antibiotic therapy for the first 2 weeks. Following 2 weeks of eradication therapy participants received TAK-438 20 mg QD along with lansoprazole matching placebo 30 mg, capsule QD for up to 6 weeks.
- Lansoprazole 30 mg: HP+ participants: Lansoprazole 30 mg, capsule, orally, BID and TAK-438 placebo-matching tablet, orally, BID along with bismuth-containing quadruple antibiotic therapy for first 2 weeks. Following 2 weeks participants received Lansoprazole 30 mg, capsule, orally, QD along with TAK-438 placebo-matching tablet, orally, QD for up to 6 weeks.
Arm/Group | TAK-438 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 75 | 73
percentage of participants | 88.0 [78.439 to 94.363] | 80.8 [69.921 to 89.099]
Statistical Analysis 1: Comparison: TAK-438 20 mg vs Lansoprazole 30 mg; Test type: Non-Inferiority — If the primary outcome measure was met, then the hypothesis for this outcome measure was that if the lower bound of the 95% CI of the difference was ≥-10%, noninferiority for TAK-438 relative to lansoprazole with regard to H pylori eradication was declared; Exact (Clopper-Pearson) = 7.2, 95% CI 2-sided [-4.469 to 18.825]

3. Secondary Outcome: Percentage of Participants With Endoscopically Confirmed Healing of GU at Week 4
Description: Endoscopic healing was defined as the disappearance of all white coats associated with GUs confirmed endoscopically.
Time Frame: Week 4
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-438 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 109 | 112
percentage of participants | 76.1 [67.035 to 83.788] | 82.1 [73.777 to 88.738]
Statistical Analysis 1: Comparison: TAK-438 20 mg vs Lansoprazole 30 mg; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Exact (Clopper-Pearson) = -6.0, 95% CI 2-sided [-16.644 to 4.741]

4. Secondary Outcome: Percentage of Participants With Post-treatment Resolution of Gastrointestinal Symptoms Associated With GU
Description: The gastrointestinal symptoms included epigastric pain [postprandial, fasting, nocturnal], abdominal bloating, nausea/vomiting, heartburn, lack of appetite. The severity of gastrointestinal symptoms associated with GU were recorded as: none = 0, mild = 1, moderate = 2 or severe = 3. The data is reported in categories for percentage of participants with resolution of gastrointestinal symptoms associated with GU.
Time Frame: Week 2 up to Week 8
Population: FAS population included all randomized participants who received at least 1 dose of the study drug. Number analyzed is the number of participants with data available for analysis for the specific category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-438 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 115 | 119
percentage of participants
  Epigastric Pain (Postprandial): number analyzed (Participants) | 19 | 25
  Epigastric Pain (Postprandial) | 78.9 [54.435 to 93.948] | 80.0 [59.296 to 93.169]
  Epigastric Pain (Fasting/Nocturnal): number analyzed (Participants) | 40 | 41
  Epigastric Pain (Fasting/Nocturnal) | 85.0 [70.165 to 94.290] | 80.5 [65.133 to 91.179]
  Abdominal Bloating: number analyzed (Participants) | 16 | 23
  Abdominal Bloating | 81.3 [54.354 to 95.953] | 65.2 [42.734 to 83.624]
  Nausea/Vomiting: number analyzed (Participants) | 9 | 8
  Nausea/Vomiting | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  Heartburn: number analyzed (Participants) | 24 | 28
  Heartburn | 95.8 [78.880 to 99.895] | 85.7 [67.335 to 95.966]
  Lack of Appetite: number analyzed (Participants) | 9 | 10
  Lack of Appetite | 77.8 [39.991 to 97.186] | 90.0 [55.498 to 99.747]
Statistical Analysis 1: Comparison: TAK-438 20 mg vs Lansoprazole 30 mg; Epigastric Pain (Postprandial); Test type: Other — [test comment as in outcome 1, analysis 1]; Exact (Clopper-Pearson) = -1.1, 95% CI 2-sided [-25.175 to 23.070]
Statistical Analysis 2: Comparison: TAK-438 20 mg; Epigastric Pain (Fasting/Nocturnal); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Exact (Clopper-Pearson) = 4.5, 95% CI 2-sided [-11.907 to 20.931]
Statistical Analysis 3: Comparison: TAK-438 20 mg vs Lansoprazole 30 mg; Abdominal Bloating; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Exact (Clopper-Pearson) = 16.0, 95% CI 2-sided [-11.255 to 43.321]
Statistical Analysis 4: Comparison: TAK-438 20 mg vs Lansoprazole 30 mg; Heartburn; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Exact (Clopper-Pearson) = 10.1, 95% CI 2-sided [-5.109 to 25.348]
Statistical Analysis 5: Comparison: TAK-438 20 mg vs Lansoprazole 30 mg; Lack of Appetite; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Exact (Clopper-Pearson) = -12.2, 95% CI 2-sided [-45.138 to 20.694]

ADVERSE EVENTS:
Time Frame: From first dose up to 4 weeks post dose (up to approximately 12 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-438 20 mg | Lansoprazole 30 mg
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/119
Serious Adverse Events (participants affected / at risk) | 3/115 | 2/119
Other Adverse Events (participants affected / at risk) | 43/115 | 15/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-438 20 mg (N=115) | Lansoprazole 30 mg (N=119)
Angina pectoris (Cardiac disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-438 20 mg (N=115) | Lansoprazole 30 mg (N=119)
Pepsinogen test positive (Investigations) | 29 | 6
Pepsinogen I increased (Investigations) | 23 | 8
Blood gastrin increased (Investigations) | 24 | 5
Alanine aminotransferase increased (Investigations) | 6 | 3
Dysgeusia (Nervous system disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT03050307/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT03050307/SAP_001.pdf